CLINICAL TRIAL: NCT05926882
Title: Efficacy of Oral Apremilast in the Treatment of Alopecia Areata at the Tertiary Care Hospital, Karachi.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr. Parisa Sanawar, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2022-GENL/321/JPMC
Record Dates: First submitted 2023-03-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apremilast tablet (Experimental): Patients will be given Oral Apremilast 30 mg twice daily after 05 days initial titration dose. The effect of treatment will be evaluated using photographs of the patients before and after the study and clinical evaluation of patients.
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 30mg — Patients will be given Oral Apremilast 30 mg twice daily after 05 days titration dose.

SUMMARY:
Alopecia areata (AA) is a disease characterized by hair cycle dysfunction and the presence of peribulbar and perifollicular mononuclear cell infiltrate.1 The majority of patients report the rapid onset of one or several well-defined, usually round, 1 to 4 cm areas of scalp hair loss. A common feature is the presence of "exclamation-mark" hairs that are broken and short hairs that taper proximally.

Commonly used treatment modalities are steroids (intra-lesional, topical or systemic), contact immunotherapy, anthraline, minoxidil, calcineurine inhibitors, topical retinoids, systemic immune modulating agents, photo-chemotherapy, dermatography wigs and hypnotherapy etc Apremilast is a newer drug. It is an oral small-molecule inhibitor of phosphodiesterase 4 (PDE4), this may be effective treatment for a variety of inflammatory skin disorders such as alopecia areata.

DETAILED DESCRIPTION:
Due to its increasing prevalence and lack of local data on its long term management, the investigators designed current study On Efficacy of Oral Apremilast in Alopecia areata in-order to evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Either gender.
* Age 20-70 years.

Exclusion Criteria:

* Patients with history of connective tissue disorder, vasculitis, seropositive and seronegative arthritis
* Patients with history of psoriasis.
* Patients excluded from the study will be patients having history of previous treatments with some systemic agents

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of Oral Apremilast in the treatment of Alopecia Areata at the Tertiary Care Hospital, Karachi | It will be assessed upto 12 weeks
  Efficacy of Oral Apremilast for 12 weeks in alopecia areata will be assessed by using SALT score ( Severity of Alopecia Tool). The SALT score is computed by measuring the percentage of hair loss in each of 4 areas of the scalp-vertex (40%), right profile (18%), left profile (18%), and posterior (24%)-and adding the total to achieve a composite score

SECONDARY OUTCOMES:
Mean difference of Salt score before and after the treatment | it will be assessed upto 12 weeks
  SALT score difference before and after the treatment will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Jabeen, FCPS, Principal Investigator — JPMC; Khadija Asadullah, FCPS, Principal Investigator — JPMC; Faiza Inam, FCPS, Principal Investigator — JPMC
Locations (1):
- JPMC, Karachi, Sindh, Pakistan